CLINICAL TRIAL: NCT06630117
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Trial to Evaluate the Safety, Tolerability, and Immunogenicity of V330 in Healthy Younger (18 to 49 Years Inclusive) and Healthy Older Participants (60 to 79 Years Inclusive).
Brief Title: A Study of V330 in Healthy Younger (18 to 49 Years Inclusive) and Healthy Older (60 to 79 Years Inclusive) Participants (V330-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: V330-001
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Dose Escalation Panel A (Experimental): Participants 18 to 49 years old will be randomized to receive V330 dose level (DL) 1 or placebo via intramuscular injection on Day 1 and Day 57.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel B (Experimental): Participants 18 to 49 years old will be randomized to receive V330 DL 3 or placebo via intramuscular injection on Day 1 and Day 57.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel C (Experimental): Participants 18 to 49 years old will be randomized to receive V330 DL 6 or placebo via intramuscular injection on Day 1 and Day 57.
  Interventions: Biological: V330; Biological: Placebo
- Dose Expansion Panel D (Experimental): Participants 18 to 49 years old will be randomized to receive a selected dose of V330 at less than or equal to DL 6 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Expansion Panel E (Experimental): Participants 18 to 49 years old will be randomized to receive a selected dose of V330 at less than or equal to DL 6 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel F (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 1 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel G (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 3 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel H (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 6 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Expansion Panel I (Experimental): Participants 60 to 79 years old will be randomized to receive a selected dose of V330 at less than or equal to DL 6 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Expansion Panel J (Experimental): Participants 60 to 79 years old will be randomized to receive a selected dose of V330 at less than or equal to DL 6 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel A1 (Experimental): Participants 18 to 49 years old will be randomized to receive V330 DL 2 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel B1 (Experimental): Participants 18 to 49 years old will be randomized to receive V330 DL 5 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel F1 (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 2 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel G1 (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 5 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo
- Dose Escalation Panel H1 (Experimental): Participants 60 to 79 years old will be randomized to receive V330 DL 4 or placebo via intramuscular injection on Day 1.
  Interventions: Biological: V330; Biological: Placebo

INTERVENTIONS:
Biological: V330 — Intramuscular injection
Biological: Placebo — Intramuscular injection

SUMMARY:
The goal of this study is to learn whether a new vaccine, V330, is safe and learn how well the body's immune system responds by making antibodies after receiving V330.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health prior to randomization
* Is an individual from 18 to 49 years of age inclusive or from 60 to 79 years of age inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of myocarditis, pericarditis, and/or myopericarditis
* Has a history of cancer

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Injection Site Adverse Events (AEs) | Up to approximately 7 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection site AEs will be recorded on a vaccination report card (VRC).
Number of Participants with Solicited Systemic AEs | Up to approximately 7 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs will be recorded on a VRC.
Number of Participants with Solicited Local AEs of Axillary Lymphadenopathy | Up to approximately 28 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Participants will be assessed for local AEs related to axillary lymphadenopathy.
Number of Participants with Immediate AEs Following Vaccinations | Up to approximately 30 minutes after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Participants will be observed following vaccination for immediate AEs.
Number of Participants with Unsolicited AEs | Up to approximately 28 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Unsolicited AEs will be recorded on a VRC.
Number of Participants with Serious AEs | Up to approximately 6 months after final vaccination
  A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event.
Number of Participants with Medically Attended Adverse Events (MAAEs) | Up to approximately 6 months after final vaccination
  A MAAE is an AE in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Routine visits are not considered MAAEs.
Number of Participants with Events of Clinical Interest (ECIs) | Up to approximately 6 months after final vaccination
  ECIs are selected serious and nonserious AEs which include but are not limited to: 1) an elevated aspartate aminotransferase or alanine aminotransferase value greater than or equal to three times the upper limit of normal (ULN) and an elevated bilirubin value of greater than two times the ULN and, at the same time, an alkaline phosphatase value of less than two times the ULN, 2) an overdose of V330.

SECONDARY OUTCOMES:
Geometric Mean Titers (GMT) of Histo-Blood Group Antigen (HBGA) Blocking Antibodies Against Vaccine-matched Norovirus (NoV) Genotypes | Up to 28 days post vaccination
  The GMT of virus like particle (VLP) serum antibody titers measured by HBGA blocking assay will be determined.
GMT of IgG Antibodies Response Against Vaccine-matched NoV Genotypes | Up to 28 days post vaccination
  The GMT of VLP serum antibody titers measured by IgG immunoassay will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0002), Glendale, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0003), Hallandale, Florida
  - Research Centers of America ( Hollywood ) ( Site 0004), Hollywood, Florida
  - QPS-MRA, LLC-Early Phase ( Site 0006), South Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com